CLINICAL TRIAL: NCT01546519
Title: A Phase Ib Open-Label Pharmacokinetics and Safety Study of the Hedgehog Pathway Inhibitor Vismodegib in Patients With Advanced Solid Malignancies Including Hepatocellular Carcinoma With Varying Degrees of Renal or Hepatic Function
Brief Title: A Study of Vismodegib in Patients With Advanced Solid Malignancies Including Hepatocellular Carcinoma With Varying Degrees of Renal or Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GP27839
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): Control cohort with normal renal and normal hepatic function
  Interventions: Drug: Vismodegib
- 2 (Experimental): Severe renal impairment and normal hepatic function
  Interventions: Drug: Vismodegib
- 3 (Experimental): Mild hepatic impairment and normal renal function
  Interventions: Drug: Vismodegib
- 4 (Experimental): Moderate hepatic impairment and normal renal function
  Interventions: Drug: Vismodegib
- 5 (Experimental): Severe hepatic impairment and normal renal function
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib — oral repeating dose of 150 mg once daily

SUMMARY:
This is a Phase Ib, open-label, multiple-center, multiple-dose study designed to evaluate the pharmacokinetics and safety of vismodegib in patients with advanced solid malignancies (including hepatocellular carcinoma and lymphoma) that are refractory to standard therapy or for whom no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed advanced solid malignancy (including hepatocellular carcinoma and lymphoma) that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Eastern Cooperative Oncology Group (ECOG) performance status </= 2 (Karnofsky >/=60%)
* Acceptable bone marrow functions
* Normal or varying degrees of renal or hepatic impairment according to NCI Organ Dysfunction Working Group criteria.
* Organ function should be stable for at least 2 weeks before Day 1. In addition, there should be no evidence of acute exacerbation of hepatic/renal disease.
* Patients with gliomas or known brain metastases who require corticosteroids or anticonvulsants must be on a stable dose of corticosteroids and seizure free for 1 month prior to enrollment. Patients with known brain metastases must be at least 4 weeks out from any radiation before starting the protocol (Day 1).
* Documented negative serum pregnancy test for women of childbearing potential
* For women of childbearing potential, agreement to the use of two acceptable methods of contraception during the study and for 7 months after discontinuation of vismodegib
* For men with female partners of childbearing potential, agreement to use a latex, non-latex, or any other male condom and to advise their female partners to use an additional acceptable method of birth control during the study and for 2 months after discontinuation of study drug
* Agreement not to donate blood/blood products during the study and for 7 months after discontinuing study drug
* For men with normal renal and hepatic function, agreement to provide semen during the vismodegib treatment period for study assessment (optional), but otherwise NOT to donate semen during the vismodegib treatment period and for 2 months after discontinuation of study drug

Exclusion Criteria:

* Pregnancy or lactation
* Chemotherapy, biologic therapy, immunotherapy, or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Investigational agents within 28 days prior to study entry (Day 1)
* Use of Pgp inhibitors within 7 days of Day 1
* Use of gastric pH altering drugs except antacids within 7 days of Day 1
* Major surgery within 14 days prior to treatment (Day 1). Patients with recent major surgery must have recovered from that surgery. Patients who are expected to have any major surgery during the study treatment period should not be enrolled.
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. History of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of vismodegib or that might affect interpretation of the results from this study or renders the patient at high risk from treatment complications.
* Severely impaired renal function (Cohort 2 only) should not have active hemolysis, and should not be on hemodialysis or peritoneal dialysis during the screening and study treatment period (Days 1-9).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (5):
- United States (5):
  - Chicago, Illinois
  - Baltimore, Maryland
  - Detroit, Michigan
  - Lebanon, New Hampshire
  - New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study with no randomization. Participants were categorized according to their baseline renal and hepatic function, and assigned to one of the five cohorts.
Pre-assignment Details: After assessing the additional data since the study initiation and after discussions with regulators, the sponsor concluded that renal impairment does not impact the pharmacokinetics of vismodegib and, therefore, a dedicated renal impairment cohort was eliminated.
Groups:
- Control Cohort With Normal Renal and Normal Hepatic Function: Participants with normal renal and normal hepatic function were included. Normal renal function was defined as Body Surface Area (BSA) - indexed creatinine clearance (CrCl) (mL/min) = / >= 60 Normal hepatic function was indicated by total bilirubin (TB) <= upper limit of normal (ULN) range and aspartate transaminase (AST) <= ULN Participants were administered 150 mg oral vismodegib once daily for 8 consecutive days (Day 1 to Day 7 doses were taken with or without food; Day 8 dose was administered on an empty stomach) at approximately the same time with about 240 mL of water.
- Mild Hepatic Impairment and Normal Renal Function (Mild HI): Participants with mild hepatic impairment and normal renal function were included.
  Mild Hepatic was defined as = TB<=ULN, AST>ULN; OR ULN<TB<=1.5× ULN, AST any Normal renal function was defined as BSA - indexed CrCl (mL/min) = / >= 60 Participants were administered 150 mg oral vismodegib once daily for 8 consecutive days (Day 1 to Day 7 doses were taken with or without food; Day 8 dose was administered on an empty stomach) at approximately the same time with about 240 mL of water.
- Moderate Hepatic Impairment and Normal Renal Function (Mod HI): Participants with moderate hepatic impairment and normal renal function were included.
  Moderate hepatic impairment was defined as 1.5 × ULN< TB<3× ULN, AST any Normal renal function was defined as BSA - indexed CrCl (mL/min) = / >= 60 Participants were administered 150 mg oral vismodegib once daily for 8 consecutive days (Day 1 to Day 7 doses were taken with or without food; Day 8 dose was administered on an empty stomach) at approximately the same time with about 240 mL of water.
- Severe Hepatic Impairment and Normal Renal Function (Sev HI): Participants with severe hepatic impairment and normal renal function were included.
  Severe hepatic impairment is defined as 3×ULN<TB<10×ULN, AST any Normal renal function was defined as BSA - indexed CrCl (mL/min) = / >= 60 Participants were administered 150 mg oral vismodegib once daily for 8 consecutive days (Day 1 to Day 7 doses were taken with or without food; Day 8 dose was administered on an empty stomach) at approximately the same time with about 240 mL of water.
Period: Overall Study
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Started | 9 | 8 | 8 | 6
Safety-Evaluable Participants | 9 | 8 | 8 | 6
Completed | 0 | 0 | 0 | 0
Not Completed | 9 | 8 | 8 | 6
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Death | 0 | 1 | 3 | 1
Not completed — related to disease progression | 2 | 2 | 2 | 1
Not completed — Physician Decision | 6 | 5 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Control Cohort With Normal Renal and Normal Hepatic Function: Participants with normal renal and normal hepatic function were included. Normal renal function was defined as Body Surface Area (BSA) - indexed creatinine clearance (CrCl) (mL/min) = / >= 60 Normal hepatic function was indicated by total bilirubin (TB) <= upper limit of normal (ULN) range and aspartate transaminase (AST) <= ULN.
  Participants were administered 150 mg oral vismodegib once daily for 8 consecutive days (Day 1 to Day 7 doses were taken with or without food; Day 8 dose was administered on an empty stomach) at approximately the same time with about 240 mL of water.
- Mild Hepatic Impairment and Normal Renal Function (Mild HI): Participants with mild hepatic impairment and normal renal function were included.
  Mild Hepatic was defined as = TB<=ULN, AST>ULN; OR ULN<TB<=1.5× ULN, AST any Normal renal function was defined as BSA - indexed CrCl (mL/min) = / >= 60. Participants were administered 150 mg oral vismodegib once daily for 8 consecutive days (Day 1 to Day 7 doses were taken with or without food; Day 8 dose was administered on an empty stomach) at approximately the same time with about 240 mL of water.
- Moderate Hepatic Impairment and Normal Renal Function (Mod HI): Participants with moderate hepatic impairment and normal renal function were included.
  Moderate hepatic impairment was defined as 1.5 × ULN< TB<3× ULN, AST any Normal renal function was defined as BSA - indexed CrCl (mL/min) = / >= 60. Participants were administered 150 mg oral vismodegib once daily for 8 consecutive days (Day 1 to Day 7 doses were taken with or without food; Day 8 dose was administered on an empty stomach) at approximately the same time with about 240 mL of water.
- Severe Hepatic Impairment and Normal Renal Function (Sev HI): Participants with severe hepatic impairment and normal renal function were included.
  Severe hepatic impairment is defined as 3×ULN<TB<10×ULN, AST any Normal renal function was defined as BSA - indexed CrCl (mL/min) = / >= 60. Participants were administered 150 mg oral vismodegib once daily for 8 consecutive days (Day 1 to Day 7 doses were taken with or without food; Day 8 dose was administered on an empty stomach) at approximately the same time with about 240 mL of water.
- Total: Total of all reporting groups
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI) | Total
Number analyzed (Participants) | 9 | 8 | 8 | 6 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (12.6) | 60.6 (14.1) | 65.8 (10.7) | 64.0 (8.4) | 63.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 2 | 1 | 7
  Male | 8 | 5 | 6 | 5 | 24

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration and Concentration at Steady-state Following Multiple Doses of Vismodegib
Description: Maximum observed plasma Concentration (Cmax) & Concentration at steady-state (Css) following multiple doses of vismodegib (150 mg QD) were analyzed. At steady state the amount of drug administered (in a given time period) is equal to the amount of drug eliminated. Blood samples for assessing Cmax and Css for analysis were collected following multiple oral doses of vismodegib at pre-dose and at 0.5, 1, 2, 4, 8 and 24 hours post-dose on Day 8. From the plasma concentration-time curve, the PK parameter Cmax and Css were determined by standard non-compartmental analysis using WinNonlin
Time Frame: Day 1,2,4 and 0, 0.5, 1, 2, 4, 8 and 24 hours post dose on Day 8
Population: Pharmacokinetic (PK) Population: A participant was considered evaluable for the PK analyses if he or she had a full profile of vismodegib samples
Measure: Mean (Standard Deviation); unit: micromolar
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Number analyzed (Participants) | 9 | 8 | 6 | 3
micromolar
  Cmax | 23.6 (9.39) | 30.7 (13.10) | 30.5 (11.60) | 20.5 (9.53)
  Css | 21.6 (9.17) | 26.9 (12.4) | 27.2 (10.5) | 19.1 (9.11)
Statistical Analysis 1: Comparison: Control Cohort With Normal Renal and Normal Hepatic Function vs Mild Hepatic Impairment and Normal Renal Function (Mild HI); Cmax Mild HI vs. Normal: Based on pooled variance estimates; Test type: Superiority or Other; Geometric mean ratio = 1.30, 90% CI 2-sided [0.95 to 1.78]
Statistical Analysis 2: Comparison: Control Cohort With Normal Renal and Normal Hepatic Function vs Moderate Hepatic Impairment and Normal Renal Function (Mod HI); Cmax Moderate HI vs. Normal: Based on pooled variance estimates; Test type: Superiority or Other; Geometric mean ratio = 1.30, 90% CI 2-sided [0.92 to 1.83]
Statistical Analysis 3: Comparison: Control Cohort With Normal Renal and Normal Hepatic Function vs Severe Hepatic Impairment and Normal Renal Function (Sev HI); Cmax Severe HI vs. Normal: Based on pooled variance estimates; Test type: Superiority or Other; Geometric mean ratio = 0.87, 90% CI 2-sided [0.55 to 1.37]
Statistical Analysis 4: Comparison: Control Cohort With Normal Renal and Normal Hepatic Function vs Mild Hepatic Impairment and Normal Renal Function (Mild HI); Css Mild HI vs. Normal: Based on pooled variance estimates; Test type: Superiority or Other; Geometric mean ratio = 1.24, 90% CI 2-sided [0.90 to 1.71]
Statistical Analysis 5: Comparison: Control Cohort With Normal Renal and Normal Hepatic Function vs Moderate Hepatic Impairment and Normal Renal Function (Mod HI); Css Moderate HI vs. Normal: Based on pooled variance estimates; Test type: Superiority or Other; Geometric mean ratio = 1.27, 90% CI 2-sided [0.89 to 1.80]
Statistical Analysis 6: Comparison: Control Cohort With Normal Renal and Normal Hepatic Function vs Severe Hepatic Impairment and Normal Renal Function (Sev HI); Css Severe HI vs. Normal: Based on pooled variance estimates; Test type: Superiority or Other; Geometric mean ratio = 0.88, 90% CI 2-sided [0.55 to 1.41]

2. Primary Outcome: The Area Under the Plasma Concentration-time Curve Over the Dosing Interval (AUC[0-24hours]) Following Multiple Doses of Vismodegib
Description: The steady state pharmacokinetic profile following oral administration of multiple doses of vismodegib included determining the area under the curve over the dosing interval (AUC[0-24 hours]). The AUC[0-24 hrs]) was determined by standard non-compartmental analysis using WinNonlin. Blood samples were collected at pre-dose and at 0.5, 1, 2, 4, 8 and 24 hours post-dose on Day 8 to estimate AUC(0-24 hrs).
Time Frame: Day 1, 2, 4 and 0, 0.5, 1, 2, 4, 8 and 24 hours postdose on Day 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Micromolar*hour
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Number analyzed (Participants) | 9 | 8 | 6 | 3
Micromolar*hour | 512 (222) | 639 (304) | 667 (274) | 437 (197)
Statistical Analysis 1: Comparison: Control Cohort With Normal Renal and Normal Hepatic Function vs Mild Hepatic Impairment and Normal Renal Function (Mild HI); AUC0-24hr Mild HI vs. Normal: Based on pooled variance estimates; Test type: Superiority or Other; Geometric mean ratio = 1.24, 90% CI 2-sided [0.89 to 1.73]
Statistical Analysis 2: Comparison: Control Cohort With Normal Renal and Normal Hepatic Function vs Moderate Hepatic Impairment and Normal Renal Function (Mod HI); AUC0-24hr Moderate HI vs. Normal: Based on pooled variance estimates; Test type: Superiority or Other; Geometric mean ratio = 1.31, 90% CI 2-sided [0.91 to 1.89]
Statistical Analysis 3: Comparison: Control Cohort With Normal Renal and Normal Hepatic Function vs Severe Hepatic Impairment and Normal Renal Function (Sev HI); AUC0-24hr Severe HI vs. Normal: Based on pooled variance estimates; Test type: Superiority or Other; Geometric mean ratio = 0.86, 90% CI 2-sided [0.53 to 1.39]

3. Secondary Outcome: The Percentage of Dose of Vismodegib in 24-hour Total Urine
Description: The percentage of dose vismodegib excreted in urine over a 24-hr total interval was estimated
Time Frame: 24 hr total interval on Day 8
Population: Pharmacokinetic (PK) Population: A participant was considered evaluable for the PK analyses if he or she had a full profile of vismodegib samples. Participants available at particular time point for assessment were included in the analysis.
Measure: Mean (Standard Deviation); unit: % Dose Excreted in 24 hr
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Number analyzed (Participants) | 8 | 7 | 3 | 3
% Dose Excreted in 24 hr | 0.792 (0.579) | 0.283 (0.253) | 0.104 (0.0485) | 0.201 (0.135)

4. Secondary Outcome: Renal Clearance of Vismodegib
Description: Renal clearance (CLR) is defined as the apparent total clearance of the drug from plasma after oral administration.
Time Frame: 0, 0.5, 1, 2, 4, 8 and 24 hours postdose on Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Number analyzed (Participants) | 8 | 7 | 3 | 3
Liter/hour | 6.76 (5.73) | 1.97 (2.24) | 0.618 (0.31) | 2.06 (1.53)

5. Secondary Outcome: Amount of Vismodegib Excreted Into Urine in 24 Hours (Ae0-24hr)
Description: The amount of total vismodegib excreted in urine over a 24-hr total interval (Ae0-24hr) was estimated.
Time Frame: 24 hr total interval on Day 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: milligrams/24 hour
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Number analyzed (Participants) | 8 | 7 | 3 | 3
milligrams/24 hour | 1.19 (0.869) | 0.425 (0.380) | 0.156 (0.0728) | 0.301 (0.203)

6. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Vismodegib
Description: Tmax is the time to reach maximum plasma concentration of vismodegib. This was a pre-specified PK parameter. However, due to minimal fluctuation of Vismodegib concentrations at steady state, this parameter could not be determined.
Time Frame: Up to 8 days
Population: PK population was the anticipated population for analysis. However, this outcome measure was not analyzed due to the minimal fluctuation of vismodegib concentrations at steady state.
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: Minimum Plasma Concentration (Cmin) of Vismodegib
Description: Cmin is defined as the minimum observed plasma concentration of Vismodegib. This was a pre-specified PK parameter. However, due to minimal fluctuation of Vismodegib concentrations at steady state, this parameter could not be determined.
Time Frame: Up to 8 days
Population: as for outcome 6
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Apparent Clearance (CL/F) of Vismodegib
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC (0-inf), expressed in liter/hour (L/hr). This was a pre-specified PK parameter. However, due to minimal fluctuation of vismodegib concentrations at steady state, this parameter could not be determined.
Time Frame: Up to 8 days
Population: as for outcome 6
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Number analyzed (Participants) | 0 | 0 | 0 | 0

9. Secondary Outcome: Apparent Non-renal Clearance (CLNR/F) of Vismodegib
Description: Apparent Non-Renal Clearance (CLNR) describes the removal of vismodegib by organs other than the kidneys. This was a pre-specified PK parameter. However, due to minimal fluctuation of vismodegib concentrations at steady state, this parameter could not be determined.
Time Frame: Up to 8 days
Population: as for outcome 6
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 60 days
Description: AEs and SAEs were collected for all the participants who received at least one dose of study medication.
Arm/Group | Control Cohort With Normal Renal and Normal Hepatic Function | Mild Hepatic Impairment and Normal Renal Function (Mild HI) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) | Severe Hepatic Impairment and Normal Renal Function (Sev HI)
Serious Adverse Events (participants affected / at risk) | 3/9 | 4/8 | 6/8 | 3/6
Other Adverse Events (participants affected / at risk) | 8/9 | 7/8 | 8/8 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Cohort With Normal Renal and Normal Hepatic Function (N=9) | Mild Hepatic Impairment and Normal Renal Function (Mild HI) (N=8) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) (N=8) | Severe Hepatic Impairment and Normal Renal Function (Sev HI) (N=6)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Pneumococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Chills (General disorders) | 1 | 0 | 0 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tumour Haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Control Cohort With Normal Renal and Normal Hepatic Function (N=9) | Mild Hepatic Impairment and Normal Renal Function (Mild HI) (N=8) | Moderate Hepatic Impairment and Normal Renal Function (Mod HI) (N=8) | Severe Hepatic Impairment and Normal Renal Function (Sev HI) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Dry eye (Eye disorders) | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 3 | 3 | 2
Vomiting (Gastrointestinal disorders) | 1 | 3 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 5 | 5 | 7 | 4
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0 | 2 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0
Waist circumference increased (Investigations) | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 3 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 1 | 2 | 2 | 2
Encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypogeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Hyposmia (Nervous system disorders) | 2 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0
Vertebral artery stenosis (Nervous system disorders) | 0 | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 0 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0
Genital lesion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 2 | 0 | 0
Venous thrombosis (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights